CLINICAL TRIAL: NCT07300423
Title: Parents' Experiences of Physical Activity in Their Children With Functional Constipation - A Qualitative Interview Study
Brief Title: Parents of Children With Constipation Will be Asked About Their Views on Their Children's Physical Activity.
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-06087-01
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Constipation - Functional
Keywords: Qualitative Research; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children with functional constipation are a large patient group that not only needs to seek care at primary healthcare centers and pediatric clinics, but many of the visits received at the emergency department are related to symptoms of constipation. The personal suffering, physically and psychologically, affects not only the child but the entire family. After the patient has started their medical treatment and received information regarding the diagnosis and dietary advice, healthcare today does not have much more to offer. The physiotherapist has currently no natural part in the team around children with constipation. Regular physical activity is recommended but lacks support in science. Physical activity has been shown to have a good effect, such as stimulating bowel movements, reducing constipation, and improving gut microbiota, in other diagnoses from the gastrointestinal tract such as irritable bowel syndrome. From a physiological perspective, physical activity is good for bowel motility; however, there is a lack of studies that can show evidence that physical activity could alleviate symptoms in functional constipation. The purpose of interviewing parents about their experiences of physical activity in their children with functional constipation is to gain a deeper understanding of physical activity in their children. Parents of 12 to15 children with functional constipation will be collected at two different pediatric clinics in Sweden to participate in the study. The method will be semistructured individual, in-depth, interviews that are transcribed verbatim and analyzed using qualitative content analysis. Both the manifest and the latent message will be analyzed. The result of this qualitative study can lead to generating new and increased knowledge about children with functional constipation and their physical activity, which can fill a knowledge gap as there is sparse previous research in the area. Knowledge from the planned study could be valuable in the long run to improve care for children with functional constipation and could lead to the physiotherapist becoming part of the team around children with functional constipation. The result from the study could also be used as a basis for future studies in the area.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 6-12 years who have functional constipation.
* Are registered at a pediatric and adolescent medicine clinic in Alingsås or Lerum due to functional constipation and are undergoing treatment for functional constipation.

Exclusion Criteria:

* Does not speak or write Swedish.
* The parent should not have impaired cognitive ability.
* The child should not have another illness/injury that could affect the ability to be physically active.
* The family should not have had the supervisor as a therapist.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parents of children with functional constipation are being recruited for the study, from two diffrent sites in western Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To explore parents' perspectives on physical activity in children suffering from functional constipation | Nov 25- April 26
  Qualitative semi structured individual in-depth interviews were analysed using qualitative content analysis. Fifteen parents of children with functional constipation are being recruited for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Närhälsan, Sörhaga Rehab, Alingsås, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dogan IG, Gursen C, Akbayrak T, Balaban YH, Vahabov C, Uzelpasaci E, Ozgul S. Abdominal Massage in Functional Chronic Constipation: A Randomized Placebo-Controlled Trial. Phys Ther. 2022 Jul 4;102(7):pzac058. doi: 10.1093/ptj/pzac058. PMID 35554601
- [Background] Bongers ME, van Wijk MP, Reitsma JB, Benninga MA. Long-term prognosis for childhood constipation: clinical outcomes in adulthood. Pediatrics. 2010 Jul;126(1):e156-62. doi: 10.1542/peds.2009-1009. Epub 2010 Jun 7. PMID 20530072
- [Background] Barberio B, Judge C, Savarino EV, Ford AC. Global prevalence of functional constipation according to the Rome criteria: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2021 Aug;6(8):638-648. doi: 10.1016/S2468-1253(21)00111-4. Epub 2021 Jun 4. PMID 34090581